CLINICAL TRIAL: NCT04043403
Title: Bilateral Closed Loop Deep Brain Stimulation for Freezing of Gait Using Neural and Kinematic Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Helen M. Bronte-Stewart, Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 52548
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will have either the Percept PC system, or Summit RC+S system from Medtronic PLC implanted.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Device: Summit RC+S (Experimental): 1. Open Loop DBS: Standard DBS therapy at a constant frequency and voltage
  2. Adaptive (Closed Loop) DBS: DBS that responds to neural or kinematic features of patient's current state
  3. Intermittent Open Loop DBS: Control for aDBS - DBS intensity or frequency changes in a manner that mimics aDBS but is pre-determined and open loop rather than being responsive to neural or kinematic signals.
  Interventions: Device: Open Loop DBS; Device: Adaptive (Closed Loop) DBS; Device: Intermittent Open Loop DBS
- Device: Percept PC (Experimental): 1. Open Loop DBS: Standard DBS therapy at a constant frequency and voltage
  2. Adaptive (Closed Loop) DBS: DBS that responds to neural features of patient's current state
  Interventions: Device: Open Loop DBS; Device: Adaptive (Closed Loop) DBS

INTERVENTIONS:
Device: Open Loop DBS — Standard DBS therapy at a constant frequency and voltage
Device: Adaptive (Closed Loop) DBS — DBS that responds to neural (Percept PC and Summit RC+S) or kinematic (Summit RC+S) features of patient's current state
Device: Intermittent Open Loop DBS — Control for aDBS - DBS intensity or frequency changes in a manner that mimics aDBS but is pre-determined and open loop rather than being responsive to neural or kinematic signals.
  Arms: Device: Summit RC+S

SUMMARY:
Deep Brain Stimulation of the subthalamic nucleus (STN) has become a standard of care, FDA-approved treatment for Parkinson's disease, with stimulation delivered at a constant amplitude and voltage, operating in an open-loop fashion that does not respond to a patient's current state. Although gait deficits and freezing of gait may initially respond to continuous open-loop deep brain stimulation (olDBS) and medication, the symptoms often recur over time.

The episodic and predictable nature of FOG makes it well suited for adaptive DBS (aDBS) and a device that overcomes the limitations of traditional high frequency olDBS and is capable of adapting therapy either in the frequency or intensity domain transiently to treat FOG while also treating other PD signs such as tremor and bradykinesia.

The purpose of this study is to determine the feasibility of an adaptive DBS system, that responds to patient-specific neural and kinematic variables with customized DBS parameters.

ELIGIBILITY:
Inclusion Criteria:

* Clinically-established PD
* Meets criteria for STN DBS eligibility as part of patient's standard medical care or already implanted in the STN with Percept(TM) PC
* The presence of complications of medication such as wearing off signs, fluctuating responses and/or dyskinesias, and/or medication refractory tremor, and/or impairment in the quality of life on or off medication due to these factors.
* Ability and willingness to return for study visits, at the initial programming and after three, six and twelve months of DBS.
* Age > 18
* Freezing of gait questionnaire (FOG-Q) score ≥ 1 and/or gait sub-score (Item 3.10) of MDS- UPDRS III ≥ 1
* Greater than or equal to 1.2 microVp between 8-35 Hz on either the LSTN or RSTN (Percept (TM) PC cohort only)

Exclusion Criteria:

* Dementia
* Untreated psychiatric disease
* Hoehn and Yahr stage 5 on or off medication (non-ambulatory)
* Age > 80
* Major surgical morbidities such as severe hypertension, coagulopathy and certain metabolic conditions that might increase the risk of hemorrhage or other surgical complications
* Presence of a cardiac pacemaker/defibrillator
* Inability to understand/sign consent
* Requires rTMS, ECT, MRI (Summit(R) RC+S cohort only), or diathermy
* Are pregnant or lactating
* Has a cranial metallic implant
* History of seizures or epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] related to Stimulation Condition | 3 Months
  A Customized Adverse Events and Tolerability Questionnaire will measure the absence/presence and frequency of paresthesias, and muscle twitching relative to each stimulation condition
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] related to quality of life | 3 Months
  The Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I, II, and IV will:
  (I) Evaluate mentation, behavior, and mood (II) Evaluate a patient's activities of daily life (IV) Measure the presence/severity of dyskinesias and other complications of therapy over time
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] related to speech | 6 Months
  The Speech Intelligibility Test (SIT) will measure changes in speech related to each stimulation condition.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] related to gait | 3 Months
  The Freezing of Gait Questionnaire (FOG-Q) will be used to record changes in gait over time

SECONDARY OUTCOMES:
Gait Parameters: Arrhythmicity | Collected up to 10 days every 3 months
  Variability in stride time during a gait task
Gait Parameters: Mean Shank Angular Velocity | Collected up to 10 days every 3 months
  Average of the peak shank angular velocities of every stride during the gait task
Gait Parameters: Mean Gait Cycle Time | Collected up to 10 days every 3 months
  Average length of time of each stride during a gait task
Percent Time Freezing | Collected up to 10 days every 3 months
  The percentage of the gait task was a participant frozen
The Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III | Collected up to 10 days every 3 months
  Portion of the scale assesses the motor signs of PD. Each item is scored on a scale from 0 (normal) to 4 (severe), with the total possible score ranging from 0 to 132.

CONTACTS AND LOCATIONS:
Overall Officials: Helen M. Bronte-Stewart, MD,MSE, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2020-06-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT04043403/ICF_000.pdf